CLINICAL TRIAL: NCT01150786
Title: Effect of Selenium Supplementation on Serum Adiponectin and Homocystein
Brief Title: Effect of Selenium on Serum Adiponectin, Homocystein and Malnutrition-inflammation Complex Syndrome in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: maryam ekramzadeh (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, maryam ekramzadeh, Ph.D, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 884746
Record Dates: First submitted 2010-06-22; First posted 2010-06-25 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Oxidative Stress; Inflammation; Malnutrition
Keywords: inflammation; oxidative stress; selenium; hemodialysis
MeSH Terms: conditions — Inflammation; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- selenium (Experimental): The patients in this arm took 200 microgram selenium yeast daily for 12 weeks.
  Interventions: Dietary Supplement: Selenium Supplement
- placebo capsule (Placebo Comparator): The patients in this arm took one placebo capsule daily for 12 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Selenium Supplement — The patients in this arm took 200 microgram selenium yeast daily for 12 weeks.
  Arms: selenium
Other: placebo — The patients in this arm took one placebo capsule daily for 12 weeks.
  Arms: placebo capsule

SUMMARY:
The aim of this study is to determine the effect of selenium supplementation as an antioxidant on serum adiponectin, HSCRP , ferritin , transferrin, albumin and homocysteine level.

DETAILED DESCRIPTION:
After screening all of 280 patients under regular HD in Faghihi Hospital Hemodialysis Center, 80 stable patients in the age range of 18-80 years old were found to be eligible for enrollment and give their informed consent to participate in this trial.The Ethics Committee of Shiraz University of Medical Sciences reviewed and approved the protocol of this study.These patients are randomly assigned in a 1:1 ratio into 2 groups of selenium(200µg) or placebo and followed for 12 weeks.Before the onset of the treatment and after the end of the treatment phase of the study, 10cc blood samples were taken from each patient. The blood was taken from the patient's arm used for hemodialysis cannulae just before the beginning of the HD session. The serum was separated by centrifugation at 3000 g/min for 5 min and stored at -70°C. Serum levels of adiponectin,high sensitive C-reactive protein (HSCRP), ferritin, transferrin, homocysteine, calcium, phosphate, albumin, blood urea nitrogen (BUN), and creatinine as well as hemoglobin (Hb) levels (g/dL) were measured in all patients at the baseline and at the end of treatment phase of study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were dialysed three times a week for at least 3 months or more

Exclusion Criteria:

* Patients who took multivitamins or immunosuppressive medications
* Patients consuming antioxidant supplements including vitamin E, vitamin C, lipoic acid, omega-3 fatty acids, soy extracts and green-tea preparations
* Patients who had active infection
* Patients who were hospitalized in the previous month.
* Being Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Subjective global Assessment(SGA)score | 12 Weeks
  change in nutritional status according to SGA from baseline to the end of intervention

SECONDARY OUTCOMES:
Serum HSCRP | 12Weeks
serum ferritin | 12Weeks
transferrin | 12 weeks
Serum adiponectin | 12Weeks
Homocystein | 12 Weeks
Serum albumin | 12Weeks
Malnutrition inflammation score(MIS) | 12 Weeks
Quality of life | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: maryam ekramzade, Ph.D, Principal Investigator — Shiraz University of Medical Sciences; moosa salehi, Ph.D, Study Director — Shiraz University of Medical Sciences; maryam ayatollahi, Ph.D, Study Chair — Shiraz University of Medical Sciences; Mohammad mahdi Sagheb, M.D, Study Chair — Shiraz University of Medical Sciences
Locations (2):
- Iran (2):
  - Shiraz University of Medical Sciences , nutrition department, Shiraz, Fars
  - Shiraz University of Medical Sciences, Shiraz, Fars